CLINICAL TRIAL: NCT04955483
Title: A Comparative Study of Virtual Single-energy Imaging and De-metallic Artifact Technology in Reducing Spinal Metallic Artifacts
Brief Title: Virtual Single-energy Imaging and De-metallic Artifact Technology in Reducing Spinal Metallic Artifacts
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018180
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2018-12

CONDITIONS: Spinal Disease
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Virtual single-energy imaging reconstruction group: Rebuild a virtual single energy map (70-140Kev, interval 10Kev)
- Virtual single energy (70-140Kev, interval 10Kev) combined with MAR reconstruction group: Rebuild a virtual single energy map (70-140Kev, interval 10Kev) combined with MAR reconstruction group
  Interventions: Diagnostic Test: Virtual single energy combined with MAR reconstruction group

INTERVENTIONS:
Diagnostic Test: Virtual single energy combined with MAR reconstruction group — combined with MAR reconstruction group
  Groups: Virtual single energy (70-140Kev, interval 10Kev) combined with MAR reconstruction group

SUMMARY:
1. Compare the effect of virtual single energy imaging and virtual single energy combined with MAR technology to remove metal artifacts in the spine. 2. Discuss the most suitable KeV of virtual single energy imaging combined with MAR technology to remove metal artifacts.

DETAILED DESCRIPTION:
The virtual single-energy imaging of energy spectrum CT combined with the metal artifact reduction technology MARS Multi Artifact Reduction System] can effectively reduce the interference of metal artifacts. This is because MAR technology corrects the image through an iterative algorithm, improves the spatial resolution, and restores the details of the adjacent tissue of the metal object. Virtual single-energy imaging technology can effectively reduce hardening artifacts. The two are used in combination to achieve the purpose of reducing metal artifacts. There have been articles about virtual single energy combined with MAR technology to reduce metal artifacts. However, the current researches mostly focus on the comparison of virtual single energy combined with MAR technology and conventional CT examination and virtual single energy imaging. There are few evaluations on the severity of metal artifacts after spinal surgery. According to different surgical methods, metal The difference in the number of implants will result in different artifact reduction effects. Secondly, the current research on the suitable KeV of virtual single energy combined with MAR technology to reduce metal artifacts is less discussed and reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery due to lumbar disc herniation or prolapse
* Patients undergoing surgical correction due to vertebral deformities.

Exclusion Criteria:

* The scan image quality caused by the patient's movement and other factors is too poor to meet the diagnostic requirements.
* Patients with only spinous processes and intervertebral spaces undergoing metal fixation after spine surgery
* Patients after spinal cord tumor surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects were selected from patients who planned to undergo routine spinal postoperative CT examinations in the radiology department from December 2018 to February 2019 in Peking University Third Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Artifact Index | 2019.2.1-2019.2.15
  Select the largest level of artifacts in the image, place a region of interest (ROI) with an area of 100-150mm2 in the soft tissue around the metal and spinal canal for CT value and standard deviation (SD) measurement, avoid the boundary area, and measure the ROI area Artifact Index ASelect the largest level of artifacts in the image, place a region of interest (ROI) with an area of 100-150mm2 in the soft tissue around the metal and spinal canal for CT value and standard deviation (SD) measurement, avoid the boundary area, and measure the ROI area Artifact Index AI

CONTACTS AND LOCATIONS:
Overall Officials: Huishu Yuan, Dr., Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No